CLINICAL TRIAL: NCT00266721
Title: Efficacy of Pancrelipase on Postprandial Belching and Bloating.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Organization: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2355
Record Dates: First submitted 2005-12-15; First posted 2005-12-19 (Estimated); Last update posted 2005-12-19 (Estimated); Status verified 2000-12

CONDITIONS: Postprandial Bloating; Postprandial Belching; Postprandial Eructation
Keywords: Pancrelipase; Abdominal bloating; Abdominal pain; Eructation
MeSH Terms: conditions — Abdominal Pain; Eructation | interventions — Pancrelipase

INTERVENTIONS:
Drug: Pancrelipase (Creon) 2 tablets with each meal

SUMMARY:
The hypothesis of this study is that the administration of pancrelipase with meals will benefit symptoms of post-prandial bloating, pain and eructation.

DETAILED DESCRIPTION:
Subjects will complete a double-blind crossover study in which, for one week periods, they will receive two pancrelipase tablets with each of the three major meals or a similarly administered identical placebo. Three times daily, subjects will rate the severity of belching, epigastric discomfort, epigastric fullness, bloating, and nausea.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have either bothersome upper abdominal discomfort, bloating (feeling of abdominal distention) or belching following meals for at least 12 month's duration. Subjects must have had a normal upper gastrointestinal endoscopy and/or upper GI series during the preceding three years.

Exclusion Criteria:

* Individuals with a history suggestive of organic disease such as recent weight loss, nausea, vomiting, GERD, recent changes in bowel habits will be excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2000-01; Study Completion 2000-10

PRIMARY OUTCOMES:
Abdominal bloating
Abdominal pain
Eructation

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Levitt, MD, Principal Investigator — Minneapolis VAMC
Locations (1):
- VAMC, Minneapolis, Minnesota, United States